CLINICAL TRIAL: NCT01015053
Title: Postoperative Pain After Pediatric Umbilical Hernia Repair: a Randomized Clinical Trial of Ultrasound-guided Bilateral Rectus Sheath Blocks Versus Local Anesthetic Infiltration
Brief Title: Postoperative Pain After Pediatric Umbilical Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Harvard Catalyst Pilot Grant (Unknown); Harvard University (Other)
Responsible Party: Principal Investigator, Catherine Chen, Attending Pediatric Surgeon, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 09-08-0398
Record Dates: First submitted 2009-11-12; First posted 2009-11-17 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Pediatric Postoperative Pain
Keywords: postoperative pain; pediatric; umbilical hernia; ropivacaine; rectus sheath block; regional block; ultrasound-guided regional block; local infiltration; ambulatory surgery
MeSH Terms: conditions — Pain, Postoperative; Hernia, Umbilical | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Regional block (Experimental): An ultrasound-guided rectus sheath block will be performed by the regional block anesthesiologist in the "regional block" arm.
  Interventions: Procedure: bilateral ultrasound-guided rectus sheath block
- Wound infiltration (Active Comparator): Local wound infiltration will be performed by the surgeon in the "wound infiltration" arm.
  Interventions: Procedure: Wound infiltration

INTERVENTIONS:
Procedure: bilateral ultrasound-guided rectus sheath block — Ultrasound is used to guide the deposition of Ropivacaine 0.2% 1cc/kg in the posterior sheath of the rectus muscle containing the peripheral nerves that innervate the abdomen.
  Other Names: ropivacaine
  Arms: Regional block
Procedure: Wound infiltration — Ropivacaine 0.2% 1cc/kg is injected subcutaneously at the site of incision by the surgeon.
  Other Names: ropivacaine
  Arms: Wound infiltration

SUMMARY:
The purpose of this study is to compare the use of ultrasound-guided bilateral rectus sheath blocks to local infiltration of anesthetic agent in the surgical wound in a pediatric population of patients undergoing umbilical hernia repair.

DETAILED DESCRIPTION:
Recent studies on adult patients' perceptions of their hospital care have shown that improvements are needed in pain management (Jha, Orav, Zheng, and Epstein). The use of regional anesthetic techniques to block specific peripheral nerves in adult patients has increased in recent decades as an alternative to general anesthesia or to decrease opioid use during and after surgery. Decreased postoperative complications have been observed, with fewer ambulatory patients requiring prolonged recovery room stays and/or costly unplanned hospital admissions (Chan, Peng, Kaszas, Middleton, Muni, Anastakis, and Graham).

Regional anesthetic techniques have not been widely performed in pediatric patients because of the challenge in requiring children to report paresthesias during needle placements. However, pediatric anesthesiologists have recently begun to use ultrasound to identify anatomy, and to guide needle insertion and local anesthetic infiltration, thereby enabling peripheral nerve blocks to be performed safely in children under general anesthesia. Several studies have illustrated that umbilical nerve blocks (Jose Maria, Götzens, and Mabrok) and rectus sheath blocks (Willschke, Bosenberg, Marhofer, Johnston, Kettner, Wanzel, and Kapral) can be used safely and effectively with ultrasound guidance in pediatric outpatient surgery. To date, few studies have explored whether ultrasound-guided regional blocks of the abdomen in children have the desired outcome of reducing postoperative pain and/or decreasing opioid use.

The use of ultrasound to guide the deposition of local anesthetic in the posterior sheath of the rectus muscle containing the peripheral nerves that innervate the abdomen may decrease postoperative pain, opioid and non-opioid analgesic consumption, as well as minimize opioid-related complications. Currently, at Children's Hospital Boston, the most common regimen for pain control after umbilical hernia repair performed under general anesthesia (i.e. standard of care) has been surgeon-administered nonspecific local anesthetic infiltration in the wound at the conclusion of surgery, followed by opioids in the Post-Anesthesia Care Unit and an oral opioid/acetaminophen combination post-discharge. In sporadic cases over the past year, several pediatric surgeons have collaborated with anesthesiologists from the pain service to allow ultrasound-guided bilateral rectus sheath blocks to be performed in patients undergoing umbilical hernia repair, usually prior to the surgical repair, and often concomitantly with surgeon-administered local anesthetic infiltration in the wound. Because of the anecdotal nature of these practices, specific conclusions regarding improvements in post-operative pain or decreased need for post-operative opioid use cannot be drawn. However, anecdotal reports from parents at the time of outpatient post-operative follow-up visits have been encouraging regarding perceived success in achieving adequate post-operative pain control in patients receiving the regional block.

We propose an interdisciplinary, prospective, randomized, single-blinded clinical trial of the use of ultrasound-guided bilateral rectus sheath blocks versus local anesthetic infiltration in a pediatric population of patients undergoing ambulatory umbilical hernia repair at Children's Hospital Boston and Children's Hospital Boston at Waltham.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who is 3 to 12 years of age
* Any patient undergoing outpatient umbilical hernia repair
* Any patient capable of expressing pain using the Faces Pain Rating Scale
* Patient has provided assent (if age 10 or older)
* Parents/guardians have provided informed consent

Exclusion Criteria:

* Any patient classified as ASA III, IV, or V by the American Society of Anesthesiologists
* Any patient with a history of Complex Regional Pain Syndrome
* Any patient with a history of chronic analgesic use
* Any patient who has used an analgesic including opioids, acetaminophen, and/or NSAID's within 24 hours prior to surgery
* Wards of the state
* Any patient with an incarcerated umbilical hernia requiring emergent surgery
* Any patient who does not speak English or Spanish
* Any patient whose primary caregiver does not speak English or Spanish
* Any patient who cannot express pain using the Faces Pain Rating Scale due to a disability
* Any patient whose primary caregiver is unable to comply with home instructions due to a disability
* Any patient less than 3 years of age or greater than 12 years of age
* Any patient with renal insufficiency
* Any patient with a bleeding disorder

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2009-11; Primary Completion 2011-05 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
postoperative pain | from emergence to 24 hrs post-discharge

SECONDARY OUTCOMES:
postoperative use of opioids and non-opioids | from emergence to 24 hrs post-discharge

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Chen, MD, MPH, Principal Investigator — Boston Children's Hospital
Locations (2):
- United States (2):
  - Children's Hospital Boston, Boston, Massachusetts
  - Children's Hospital Boston at Waltham, Waltham, Massachusetts

REFERENCES:
- [Background] Jha AK, Orav EJ, Zheng J, Epstein AM. Patients' perception of hospital care in the United States. N Engl J Med. 2008 Oct 30;359(18):1921-31. doi: 10.1056/NEJMsa0804116. PMID 18971493
- [Background] Chan VW, Peng PW, Kaszas Z, Middleton WJ, Muni R, Anastakis DG, Graham BA. A comparative study of general anesthesia, intravenous regional anesthesia, and axillary block for outpatient hand surgery: clinical outcome and cost analysis. Anesth Analg. 2001 Nov;93(5):1181-4. doi: 10.1097/00000539-200111000-00025. PMID 11682392
- [Background] de Jose Maria B, Gotzens V, Mabrok M. Ultrasound-guided umbilical nerve block in children: a brief description of a new approach. Paediatr Anaesth. 2007 Jan;17(1):44-50. doi: 10.1111/j.1460-9592.2006.02025.x. PMID 17184431
- [Background] Willschke H, Bosenberg A, Marhofer P, Johnston S, Kettner SC, Wanzel O, Kapral S. Ultrasonography-guided rectus sheath block in paediatric anaesthesia--a new approach to an old technique. Br J Anaesth. 2006 Aug;97(2):244-9. doi: 10.1093/bja/ael143. Epub 2006 Jun 23. PMID 16798774
- [Derived] Dingeman RS, Barus LM, Chung HK, Clendenin DJ, Lee CS, Tracy S, Johnson VM, Dennett KV, Zurakowski D, Chen C. Ultrasonography-guided bilateral rectus sheath block vs local anesthetic infiltration after pediatric umbilical hernia repair: a prospective randomized clinical trial. JAMA Surg. 2013 Aug;148(8):707-13. doi: 10.1001/jamasurg.2013.1442. PMID 23760519